CLINICAL TRIAL: NCT05041530
Title: A Prospective, Multi-Center, Single Arm, Feasibility Study Using REBUILD Bioabsorbable™ for Closure of the Abdominal Wall After Oncologic Laparotomy
Brief Title: Abdominal Wall Closure After Laparotomy in Oncologic Surgery
Acronym: REBUILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AbSolutions Med Inc. (Industry)
Collaborators: Cogent Technologies Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-0001
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Laparotomy
Keywords: Laparotomy; Abdominal Wall Closure

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, single-arm, feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- REBUILD (Experimental): Subjects who meet the inclusion criteria and agree to participate in the study will be enrolled and undergo oncologic laparotomy per the standard of care. The abdominal wall will be closed with REBUILD Bioabsorbable and suture of the surgeon's choice.
  Interventions: Device: REBUILD Bioabsorbable

INTERVENTIONS:
Device: REBUILD Bioabsorbable — REBUILD is an investigational medical device designed to be used with third-party suture to distribute suture tension in abdominal wall closures.

SUMMARY:
The REBUILD Study is a first-in-human evaluation of the safety and performance of REBUILD Bioabsorbable.

DETAILED DESCRIPTION:
REBUILD is an investigational medical device designed to be used with third-party suture to distribute suture tension in abdominal wall closures. In this study, REBUILD will be used in oncology patients undergoing an open, elective, intent-to-cure, laparotomy procedure. The study is a prospective, non-randomized, multi-center study designed to generate descriptive data about the use of REBUILD. The primary safety outcome is reported device-related adverse events. The primary performance outcome is the integrity of the abdominal wall over one year assessed by clinical examination of the abdomen. If available, CT studies performed within 12 months post-procedure will be used to confirm apposition of the medial border of the rectus muscles and integrity of the abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18-75 years of age
2. Patient is scheduled for oncologic, open, elective, intent-to-cure laparotomy
3. Patient is able to provide written informed consent
4. Patient is able and willing to comply with all study requirements

Exclusion Criteria:

1. Patient is scheduled for a palliative procedure
2. Patient has had previous failed surgical repair of a ventral or incisional hernia
3. Patient has a current infection at the intended surgical site
4. Patient is participating in a concurrent investigational medical device study
5. Patient is pregnant or planning on becoming pregnant during the study period
6. Patient has a history of psychological condition, drug or alcohol misuse which may interfere with their ability to be compliant with post-operative visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  The number of device-related adverse events
Performance | 12 months
  The number of subjects with abdominal wall integrity at 3-, 6-, and 12-months post-surgery. Abdominal wall integrity will be assessed via clinical examination of the abdomen to identify a fascial defect, bulge, reducible palpable mass, or discomfort with a cough impulse. Standard of care CT or MR imaging that is performed within 12 months of the surgery will be evaluated to confirm apposition of the medial border of the rectus abdominis muscles and integrity of the abdominal wall.

CONTACTS AND LOCATIONS:
Overall Officials: Luis J Palacios Fuenmayor, MD, Principal Investigator — Clinica Las Americas
Locations (2):
- Colombia (2):
  - Clinica Medellin, Medellín, Antioquia
  - Clinica Las Americas, Medellín

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kokotovic D, Bisgaard T, Helgstrand F. Long-term Recurrence and Complications Associated With Elective Incisional Hernia Repair. JAMA. 2016 Oct 18;316(15):1575-1582. doi: 10.1001/jama.2016.15217. PMID 27750295
- [Background] Flum DR, Horvath K, Koepsell T. Have outcomes of incisional hernia repair improved with time? A population-based analysis. Ann Surg. 2003 Jan;237(1):129-35. doi: 10.1097/00000658-200301000-00018. PMID 12496540
- [Background] Hawn MT, Snyder CW, Graham LA, Gray SH, Finan KR, Vick CC. Long-term follow-up of technical outcomes for incisional hernia repair. J Am Coll Surg. 2010 May;210(5):648-55, 655-7. doi: 10.1016/j.jamcollsurg.2009.12.038. PMID 20421023
- [Background] Deeken CR, Matthews BD. Characterization of the Mechanical Strength, Resorption Properties, and Histologic Characteristics of a Fully Absorbable Material (Poly-4-hydroxybutyrate-PHASIX Mesh) in a Porcine Model of Hernia Repair. ISRN Surg. 2013 May 28;2013:238067. doi: 10.1155/2013/238067. Print 2013. PMID 23781348
- [Background] Glauser PM, Brosi P, Speich B, Kaser SA, Heigl A, Rosenberg R, Maurer CA. Prophylactic Intraperitoneal Onlay Mesh Following Midline Laparotomy-Long-Term Results of a Randomized Controlled Trial. World J Surg. 2019 Jul;43(7):1669-1675. doi: 10.1007/s00268-019-04964-6. PMID 30824961
- [Background] Kohler A, Lavanchy JL, Lenoir U, Kurmann A, Candinas D, Beldi G. Effectiveness of Prophylactic Intraperitoneal Mesh Implantation for Prevention of Incisional Hernia in Patients Undergoing Open Abdominal Surgery: A Randomized Clinical Trial. JAMA Surg. 2019 Feb 1;154(2):109-115. doi: 10.1001/jamasurg.2018.4221. PMID 30476940
- [Background] San Miguel C, Melero D, Jimenez E, Lopez P, Robin A, Blazquez LA, Lopez-Monclus J, Gonzalez E, Jimenez C, Garcia-Urena MA. Long-term outcomes after prophylactic use of onlay mesh in midline laparotomy. Hernia. 2018 Dec;22(6):1113-1122. doi: 10.1007/s10029-018-1833-x. Epub 2018 Oct 4. PMID 30288617
- [Background] Jairam AP, Timmermans L, Eker HH, Pierik REGJM, van Klaveren D, Steyerberg EW, Timman R, van der Ham AC, Dawson I, Charbon JA, Schuhmacher C, Mihaljevic A, Izbicki JR, Fikatas P, Knebel P, Fortelny RH, Kleinrensink GJ, Lange JF, Jeekel HJ; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement versus primary suture only in midline laparotomies (PRIMA): 2-year follow-up of a multicentre, double-blind, randomised controlled trial. Lancet. 2017 Aug 5;390(10094):567-576. doi: 10.1016/S0140-6736(17)31332-6. Epub 2017 Jun 20. PMID 28641875
- [Background] Muysoms FE, Detry O, Vierendeels T, Huyghe M, Miserez M, Ruppert M, Tollens T, Defraigne JO, Berrevoet F. Prevention of Incisional Hernias by Prophylactic Mesh-augmented Reinforcement of Midline Laparotomies for Abdominal Aortic Aneurysm Treatment: A Randomized Controlled Trial. Ann Surg. 2016 Apr;263(4):638-45. doi: 10.1097/SLA.0000000000001369. PMID 26943336
- [Background] Bali C, Papakostas J, Georgiou G, Kouvelos G, Avgos S, Arnaoutoglou E, Papadopoulos G, Matsagkas M. A comparative study of sutured versus bovine pericardium mesh abdominal closure after open abdominal aortic aneurysm repair. Hernia. 2015 Apr;19(2):267-71. doi: 10.1007/s10029-014-1262-4. Epub 2014 May 13. PMID 24820007
- [Background] Deerenberg EB, Harlaar JJ, Steyerberg EW, Lont HE, van Doorn HC, Heisterkamp J, Wijnhoven BP, Schouten WR, Cense HA, Stockmann HB, Berends FJ, Dijkhuizen FPH, Dwarkasing RS, Jairam AP, van Ramshorst GH, Kleinrensink GJ, Jeekel J, Lange JF. Small bites versus large bites for closure of abdominal midline incisions (STITCH): a double-blind, multicentre, randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1254-1260. doi: 10.1016/S0140-6736(15)60459-7. Epub 2015 Jul 15. PMID 26188742
- [Background] Garcia-Urena MA, Lopez-Monclus J, Hernando LA, Montes DM, Valle de Lersundi AR, Pavon CC, Ceinos CJ, Quindos PL. Randomized controlled trial of the use of a large-pore polypropylene mesh to prevent incisional hernia in colorectal surgery. Ann Surg. 2015 May;261(5):876-81. doi: 10.1097/SLA.0000000000001116. PMID 25575254
- [Background] Sarr MG, Hutcher NE, Snyder S, Hodde J, Carmody B. A prospective, randomized, multicenter trial of Surgisis Gold, a biologic prosthetic, as a sublay reinforcement of the fascial closure after open bariatric surgery. Surgery. 2014 Oct;156(4):902-8. doi: 10.1016/j.surg.2014.06.022. PMID 25239343
- [Background] Khorgami Z, Shoar S, Laghaie B, Aminian A, Hosseini Araghi N, Soroush A. Prophylactic retention sutures in midline laparotomy in high-risk patients for wound dehiscence: a randomized controlled trial. J Surg Res. 2013 Apr;180(2):238-43. doi: 10.1016/j.jss.2012.05.012. Epub 2012 May 24. PMID 22677612
- [Background] Curro G, Centorrino T, Low V, Sarra G, Navarra G. Long-term outcome with the prophylactic use of polypropylene mesh in morbidly obese patients undergoing biliopancreatic diversion. Obes Surg. 2012 Feb;22(2):279-82. doi: 10.1007/s11695-011-0486-y. PMID 21809056
- [Background] Rasic Z, Schwarz D, Adam VN, Sever M, Lojo N, Rasic D, Matejic T. Efficacy of antimicrobial triclosan-coated polyglactin 910 (Vicryl* Plus) suture for closure of the abdominal wall after colorectal surgery. Coll Antropol. 2011 Jun;35(2):439-43. PMID 21755716
- [Background] Bloemen A, van Dooren P, Huizinga BF, Hoofwijk AG. Randomized clinical trial comparing polypropylene or polydioxanone for midline abdominal wall closure. Br J Surg. 2011 May;98(5):633-9. doi: 10.1002/bjs.7398. Epub 2011 Jan 19. PMID 21254041
- [Background] Bevis PM, Windhaber RA, Lear PA, Poskitt KR, Earnshaw JJ, Mitchell DC. Randomized clinical trial of mesh versus sutured wound closure after open abdominal aortic aneurysm surgery. Br J Surg. 2010 Oct;97(10):1497-502. doi: 10.1002/bjs.7137. PMID 20603858
- [Background] El-Khadrawy OH, Moussa G, Mansour O, Hashish MS. Prophylactic prosthetic reinforcement of midline abdominal incisions in high-risk patients. Hernia. 2009 Jun;13(3):267-74. doi: 10.1007/s10029-009-0484-3. Epub 2009 Mar 5. PMID 19262985
- [Background] Henriksen NA, Deerenberg EB, Venclauskas L, Fortelny RH, Miserez M, Muysoms FE. Meta-analysis on Materials and Techniques for Laparotomy Closure: The MATCH Review. World J Surg. 2018 Jun;42(6):1666-1678. doi: 10.1007/s00268-017-4393-9. PMID 29322212
- [Background] Taylor DA, Merten SL, Sandercoe GD, Gahankari D, Ingram SB, Moncrieff NJ, Ho K, Sellars GD, Magnusson MR. Abdominoplasty Improves Low Back Pain and Urinary Incontinence. Plast Reconstr Surg. 2018 Mar;141(3):637-645. doi: 10.1097/PRS.0000000000004100. PMID 29481394
- [Background] Nenshi R, Bensimon C, Wood T, Wright F, Smith AJ, Brenneman F. Complex abdominal wall hernias as a barrier to quality of life in cancer survivors. Can J Surg. 2019 Mar 22;62(3):1-7. doi: 10.1503/cjs.014917. Online ahead of print. PMID 30900432
- [Background] Burger JW, Lange JF, Halm JA, Kleinrensink GJ, Jeekel H. Incisional hernia: early complication of abdominal surgery. World J Surg. 2005 Dec;29(12):1608-13. doi: 10.1007/s00268-005-7929-3. PMID 16311846
- [Background] Harlaar JJ, Deerenberg EB, Dwarkasing RS, Kamperman AM, Kleinrensink GJ, Jeekel J, Lange JF. Development of incisional herniation after midline laparotomy. BJS Open. 2017 May 10;1(1):18-23. doi: 10.1002/bjs5.3. eCollection 2017 Feb. PMID 29951601
- [Background] Onyekwelu I, Yakkanti R, Protzer L, Pinkston CM, Tucker C, Seligson D. Surgical Wound Classification and Surgical Site Infections in the Orthopaedic Patient. J Am Acad Orthop Surg Glob Res Rev. 2017 Jun 13;1(3):e022. doi: 10.5435/JAAOSGlobal-D-17-00022. eCollection 2017 Jun. PMID 30211353
- [Background] Playforth MJ, Sauven PD, Evans M, Pollock AV. The prediction of incisional hernias by radio-opaque markers. Ann R Coll Surg Engl. 1986 Mar;68(2):82-4. PMID 3954314
- [Background] Pollock AV, Evans M. Early prediction of late incisional hernias. Br J Surg. 1989 Sep;76(9):953-4. doi: 10.1002/bjs.1800760926. No abstract available. PMID 2804595
- See also: American Society of Anesthesiologists Physical Status Classification System — https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system